CLINICAL TRIAL: NCT03093103
Title: Effects of the SGLT2 Inhibitor Empagliflozin on Renal Tissue Oxygenation in Non-diabetic Subjects
Brief Title: Empagliflozin and Renal Oxygenation in Healthy Volunteers
Acronym: EMPA-REIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Michel Burnier, Professor, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2016-00099
Record Dates: First submitted 2017-03-16; First posted 2017-03-28 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Nephropathy
Keywords: empagliflozin; kidney; BOLD-MRI
MeSH Terms: conditions — Kidney Diseases | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: Randomised placebo-controlled double blind trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Placebo and Empagliflozin pills
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- empagliflozin 10mg (Active Comparator): Empagliflozin (Jardiance) 10mg is an SGLT-2inhibitor. The drug will be taken qd for 4 weeks.
  Interventions: Drug: Empagliflozin 10 mg
- Placebo (Placebo Comparator): Placebo will be taken qd for 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin 10 mg — Prescription of empagliflozin 10 mg once a day Follow-up of renal parameters including BOLD MRI
  Other Names: Jardiance
  Arms: empagliflozin 10mg
Drug: Placebo — Prescription of a placebo once a day Follow-up of renal parameters including BOLD MRI
  Arms: Placebo

SUMMARY:
SGLT-2 inhibitors belong to a new class of hypoglycemic drugs with the unique property of decreasing blood glucose through an increase in glucosuria. These drugs inhibit the sodium glucose transporter 2 (SGLT2) expressed at the luminal membrane of the proximal tubule.

SGLT-2 inhibition in type 2 diabetic subjects and in healthy volunteers shifts the threshold for renal glucose excretion to lower levels. This effect is independent from insulin. The inhibition of SGLT2 decreases HbA1C, systolic blood pressure and weight in diabetic subjects. Recently, the EMPA-REG trial demonstrated a decrease in cardiovascular mortality and renal endpoints in empagliflozin treated type 2 diabetic patients with established cardio-vascular disease.

Because this novel hypoglycemic drug has unique and direct effects on renal tissue metabolism, it is important to better examine its effects on the kidney. With this study, we propose to explore the effects of empagliflozin on renal tissue oxygenation. Our hypothesis is that SGLT-2 inhibition decreases renal cortical energy requirements with consequently an increase in renal tissue oxygenation.

DETAILED DESCRIPTION:
This study is a double-blind, randomized, placebo-controlled study that will examine the acute and chronic renal effects of empagliflozin in healthy volunteers.

A total of 45 healthy volunteers will be included in the study: 15 normal weight, 15 overweight (BMI: 25-30kg/m2) and 15 obese (BMI>30kg/m2) non diabetic subjects (as determined after an oral glucose tolerance test).

Empagliflozin 10mg vs placebo will be administered in a blinded fashion qd. The acute and chronic renal response to empagliflozin will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Normal weight (BMI: 19-24.9kg/m2), overweight (BMI:25-30kg/m2) or obesity (BMI>30kg/m2)
* Men and women (with a negative pregnancy test) during the follicular phase of the menstrual cycle. All groups will have a balanced number of men and women.
* OGTT/HbA1C: normal or pre-diabetes
* eGFR>60ml/min, albumin/creatinine ratio <3.3mg/mmol (<30 mg/g)
* Signed consent form
* Normal renal ultrasound
* Normal urine dipstick

Exclusion Criteria:

* Antihypertensive therapy
* NSAID treatment
* Former bariatric surgery
* Age<18y or >50y
* At risk of dehydration or hypotension
* Past history of recurrent genital or urinary tract infections
* Contra-indication for MR imaging (pacemaker or other implanted metallic device, claustrophobia)
* Pregnancy
* Sustained systolic blood pressure >150mmHg or diastolic blood pressure >95mmHg

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2017-03-16 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Renal oxygenation | 18 months
  The acute and chronic effect of empagliflozin on renal oxygenation will be assessed by BOLD-MRI

SECONDARY OUTCOMES:
Acute and chronic effects of empagliflozin on diurnal and nocturnal sodium, potassium, uric acid, calcium, phosphate, glucose and lithium clearances after 4 weeks treatment | 18 months
  Will be assessed on 24h urinary collections
Acute and chronic effects of empagliflozin on renal resistance indexes and renal volume after 4 weeks treatment | 18 months
  Will be assessed by renal ultrasound
Effects of empagliflozin on 24h blood pressure mesaurements | 18 months
  WIll be assessed by ambulatory blood pressure measurements
Effect of body weight on the renal response to empagliflozin | 18 months
  Different groups of BMI will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Michel Burnier, Prof, Principal Investigator — Service de Néphrologie CHUV
Locations (1):
- Service de Néphrologie, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zanchi A, Pruijm M, Muller ME, Ghajarzadeh-Wurzner A, Maillard M, Dufour N, Bonny O, Wuerzner G, Burnier M. Twenty-Four Hour Blood Pressure Response to Empagliflozin and Its Determinants in Normotensive Non-diabetic Subjects. Front Cardiovasc Med. 2022 Mar 22;9:854230. doi: 10.3389/fcvm.2022.854230. eCollection 2022. PMID 35391843
- [Derived] Harmacek D, Pruijm M, Burnier M, Muller ME, Ghajarzadeh-Wurzner A, Bonny O, Zanchi A. Empagliflozin Changes Urine Supersaturation by Decreasing pH and Increasing Citrate. J Am Soc Nephrol. 2022 Jun;33(6):1073-1075. doi: 10.1681/ASN.2021111515. Epub 2022 Apr 6. PMID 35387874
- [Derived] Zanchi A, Burnier M, Muller ME, Ghajarzadeh-Wurzner A, Maillard M, Loncle N, Milani B, Dufour N, Bonny O, Pruijm M. Acute and Chronic Effects of SGLT2 Inhibitor Empagliflozin on Renal Oxygenation and Blood Pressure Control in Nondiabetic Normotensive Subjects: A Randomized, Placebo-Controlled Trial. J Am Heart Assoc. 2020 Jul 7;9(13):e016173. doi: 10.1161/JAHA.119.016173. Epub 2020 Jun 20. PMID 32567439
- [Derived] Muller ME, Pruijm M, Bonny O, Burnier M, Zanchi A. Effects of the SGLT-2 Inhibitor Empagliflozin on Renal Tissue Oxygenation in Non-Diabetic Subjects: A Randomized, Double-Blind, Placebo-Controlled Study Protocol. Adv Ther. 2018 Jun;35(6):875-885. doi: 10.1007/s12325-018-0708-y. Epub 2018 May 25. PMID 29802538